CLINICAL TRIAL: NCT01330251
Title: Laihdutusleikkauksen Vaikutus Diabetekseen
Brief Title: The Effect of Gastric Bypass Surgery on Diabetes
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Laihdutusleikkaustutkimus
Record Dates: First submitted 2011-03-22; First posted 2011-04-06 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, feces, intestinal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with diabetes having Roux-en-Y gastric bypass
- Patients without diabetes having Roux-en-Y gastric bypass
- Control subjects (patients having gastroscopy, no surgery)

SUMMARY:
This study will investigate the effects of gastric bypass surgery on type II diabetes. The study will recruit patients with type II diabetes having Roux-en-Y gastric bypass, patients without type II diabetes having Roux-en-Y gastric bypass, and control subjects (patients having gastroscopy, but no surgery). Targeted enrollment is 30 patients per group. Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy. Meal test with incretin measurements, and feces and blood samplings are performed before and after surgery

Hypotheses are:

* The pathogenesis of type II diabetes is linked to changes in the expression of intestinal endocrine cells
* The changes in the incretine excretion after the gastric bypass surgery partly explain the amelioration of type II diabetes
* The oxidation of lipoprotein is diminished after the gastric bypass surgery slowing the development of atherosclerosis
* The immunologic functions of the intestine are changed by the gastric bypass surgery attenuating systemic inflammation
* The gastric bypass surgery changes cholesterol and bile acid metabolism
* The gastric bypass surgery changes the fecal microbiota

Primary end points are:

* Changes in the amounts of endocrine cells in ventricle, duodenum and jejunum
* Changes in the incretine secretion studied with liquid meal test
* Changes in the oxidation of lipoproteins
* Changes in the immunologic markers in ventricle, duodenum and jejunum
* Changes in the amounts of phytosterols, cholesterol metabolites and bile acids
* Changes in fecal microbiota

ELIGIBILITY:
Inclusion Criteria (patients with surgery):

* Patients having Roux-en-Y gastric bypass (according to clinical guidelines)
* Age: 18-65 years

Inclusion Criteria (control patients without surgery):

* Patients having gastroscopy (for various clinical reasons)

Exclusion Criteria:

* Diabetes (applies for control patients)
* BMI over 30 (applies for control patients)
* Insulin treatment
* Oral corticosteroid treatment
* Chronic inflammatory disease
* Coeliac disease
* Malignant disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are recruited from Oulu University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in the amounts of endocrine cells in ventricle, duodenum and jejunum | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy
Changes in the incretine secretion studied with liquid meal test | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy
Changes in the oxidation of lipoproteins | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy
Changes in the immunologic markers in ventricle, duodenum and jejunum | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy
Changes in the amounts of phytosterols, cholesterol metabolites and bile acids | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy
Changes in fecal microbiota | baseline to 6 months
  Samples of intestine are taken prior to surgery in gastroscopy, during surgery, and 6 months after surgery during gastroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Vesa Koivukangas, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Zhao S, Horkko S, Savolainen MJ, Koivukangas V, Makinen VP, Ala-Korpela M, Hukkanen J. Short-Term Metabolic Changes and Their Physiological Mediators in the Roux-en-Y Gastric Bypass Bariatric Surgery. Obes Surg. 2024 Feb;34(2):625-634. doi: 10.1007/s11695-023-07042-y. Epub 2024 Jan 9. PMID 38191968
- [Derived] Rahunen R, Kummu O, Koivukangas V, Hautajarvi H, Hakkola J, Rysa J, Hukkanen J. Pregnane X Receptor-4beta-Hydroxycholesterol Axis in the Regulation of Overweight- and Obesity-Induced Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e023492. doi: 10.1161/JAHA.121.023492. Epub 2022 Mar 1. PMID 35229613